CLINICAL TRIAL: NCT05211206
Title: Association Between Peri-procedural Intravenous Hydration and Post- Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Brief Title: IV Fluids and Post-ERCP Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: McGill University (Other); University of Ottawa (Other); Queen's University (Other); Halton Health (Oakville) (Unknown); Island Health, Victoria, BC (Other)
Responsible Party: Sponsor
Other Study IDs: REB21-1885
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: ERCP
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aggressive hydration: Patients with greater than or equal to 2 L of intravenous crystalloid fluids administered within the immediate pre-, peri- and post-procedural period
  Interventions: Other: IV fluids
- Conservative hydration: Patients with less than 1 L of intravenous crystalloid fluids administered within the immediate pre-, peri- and post-procedural period
  Interventions: Other: IV fluids

INTERVENTIONS:
Other: IV fluids — Amount of intravenous fluids delivered

SUMMARY:
Aggressive intravenous hydration has been shown in randomized trials to prevent post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (PEP), though studied regimens are often impractical. To date, no studies have prospectively assessed short-term (60-90 minute) aggressive hydration regimens that are feasible for outpatients undergoing ERCP and subsequent discharge. Furthermore, little is known with regard to fluid type, volume, and timing with respect to ERCP. In this study, we will aim to assess whether the amount of peri-procedural intravenous fluid administered around the time of ERCP is associated with the risk of PEP (the primary outcome).

DETAILED DESCRIPTION:
1. Background and Rationale

   While very effective, endoscopic retrograde cholangiopancreatography (ERCP) is widely known to have the highest adverse event (AE) profile among all commonly performed endoscopic procedures, with a collective AE rate of >10%. Common AEs include post-ERCP pancreatitis (PEP), bleeding, cholangitis, cholecystitis, perforation, and cardiopulmonary events. PEP is the most common, with estimated rates of 5-10%. It is noteworthy that both the incidence of PEP and its associated mortality are rising.

   It is of critical priority to patients, practitioners, and health administrators to investigate factors associated with all AEs and unplanned healthcare encounters (UHEs) following ERCP, especially given that most ERCPs are performed on an outpatient basis. The per-admission costs of post-ERCP UHEs are substantial, exceeding $10,000 and $70,000 for pancreatitis and cholangitis, respectively. PEP alone accounts for an estimated $200+ million in annual healthcare spending in the United States. Thus, researchers must prioritize the study of ERCP outcomes, striving to both identify and modify factors leading to AEs and UHEs.

   Peri-procedural fluid management and its relationship with ERCP outcomes also remains incompletely understood. Aggressive intravenous hydration (AH) has been shown to reduce the risk of PEP compared with standard peri-procedural hydration regimens. However, all AH regimens studied to date involve continuous hydration for 8-24 hours, which is impractical and thus non-generalizable to almost all North American outpatient ERCPs practices. To date, no studies have prospectively assessed short-term (60-90 minute) aggressive hydration regimens that are feasible for outpatients undergoing ERCP and subsequent discharge. Furthermore, little is known with regard to fluid type, volume, and timing with respect to ERCP.
2. Research Question and Objectives

   In this study, we will aim to assess whether the amount of peri-procedural intravenous fluid administered around the time of ERCP is associated with the risk of PEP (the primary outcome).
3. Methods

Design: This is a retrospective cohort study where all data used to answer the proposed research question will be obtained from research data previously collected under REB18-0410. REB18-0410 (CReATE) is a multicenter prospective cohort study that recruits patients undergoing ERCP during which various relevant clinical and patient demographic data have been collected. The objective of REB18-0410 is to determine the clinical effectiveness and adverse event profile of ERCP.

The exposure variable for this study will be a the total peri-procedural IV fluid volume administered, measured and reported as a continuous variable. In addition to these variables, other parameters we will assess include: the presence and timing of pharmacologic PEP prophylaxis, extent and timing of trainee involvement, the number and timing of common bile duct (CBD) cannulation attempts, the depth, timing, trajectory and number of PD cannulation(s), the presence and extent of PD opacification, the size(s) of sphincterotomy and/or sphincteroplasty, intra-procedural pathology, and the composition, caliber and length of any PD or CBD stent(s).

Outcomes: The primary outcome will be PEP, using established definitions. Secondary outcomes (defined a priori) will include PEP severity, overall and specific AEs (bleeding, cholangitis, cardio-pulmonary events), cannulation time and success rate, as well as overall procedure time and success rate.

Sample Size and Power: Using a cutoff of a total peri-procedural IV fluid volume of ≥ 2 L (versus < 1 L), a minimum of 1,530 patients are anticipated to meet the exposure definition, with an anticipated 12,750 patients that will meet the control definition. We will be able to demonstrate increases in PEP risk from 5.0% to 6.8% (a relative increase of 36%) with 82.3% power or from 5.0% to 7.0% (a relative increase of 40%) with 88.6% power.

Statistical Analysis: Variables will be compared using Student's t-test for measured variables and chi-squared test for categorical variables. P values < 0.05 will be considered significant. We will use multivariable logistic regression to assess associations between risk factors and having PEP versus not having PEP. Clinically relevant subgroup analyses will also be performed by relevant patient-, endoscopist-, and procedure-related characteristics. Odds ratios per outcome will be reported with 95% CIs.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred for ERCP, regardless of indication;
* Subject age 18 years or older;
* Subject able to give informed consent to involvement be included.

Exclusion Criteria:

* Subject has a standard contraindication to ERCP;
* Subject or surrogate unable or unwilling to provide informed consent;
* Subject age < 18 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred to a hospital-based endoscopy unit for consideration of ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
post-ERCP pancreatitis | 30 days
  Number of participants with any 2 of: (1) epigastric abdominal pain, (2) serum amylase/lipase >3x the upper limit of normal, (3) imaging findings consistent with acute pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Nauzer Forbes, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- Peter Lougheed Hospital, Calgary, Alberta, Canada